CLINICAL TRIAL: NCT02588248
Title: L-Menthol Injection as a Novel Technique During Colonoscopy: The MINT-C Study
Brief Title: L-Menthol Injection as a Novel Technique During Colonoscopy
Acronym: MINT-C
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor/Investigator has decided to close out the study
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Richard C. K. Wong, MD., M.D., University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 05-15-07
Record Dates: First submitted 2015-10-06; First posted 2015-10-27 (Estimated); Results first posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-03

CONDITIONS: Colonic Polyps; Colon Cancer
Keywords: Colon Cancer; Colonic Polyps; L-Menthol; C-Mint
MeSH Terms: conditions — Colonic Polyps; Colonic Neoplasms | interventions — peppermint oil; Menthol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peppermint Oil (Experimental): Solution A) Peppermint oil solution (1.6% peppermint oil, which is 0.8% L-menthol)
  Ingredients:
  1. 16mL of peppermint oil (provided by the NowFoods® company)
  2. 0.4mL of Tween® 80 (i.e. Polysorbate 80) - this is a commonly used food additive that acts as a surfactant to bring the peppermint oil into solution
  3. 1L prepackage sterile water
  4. 2.6mL of undyed simethicone
  Interventions: Drug: Peppermint Oil
- Placebo (Placebo Comparator): Solution B) Placebo solution
  Ingredients:
  1. 0.4mL of Tween® 80 (i.e. Polysorbate 80) - this is a commonly used food additive that acts as a surfactant to bring the peppermint oil into solution
  2. 1L prepackage sterile water
  3. 2.6mL of undyed simethicone
     Instructions to prepare:
  4. Add tween and simethicone to sterile water. Then, shake vigorously.
  5. Once solution has settled, and patient has been randomized, draw 20mL of solution into a plastic syringe
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Peppermint Oil — During the colonoscopy the Endoscopists will be required to deliver intraluminally 1 syringe at the cecum and 1 syringe in the sigmoid colon. Up to 2 additional doses can be delivered at the discretion of the endoscopist up to a maximum of 4 total doses (max total dose = 640 mg of L-Menthol).
  Other Names: L-Menthol
  Arms: Peppermint Oil
Other: Placebo — During the colonoscopy the Endoscopists will be required to deliver intraluminally 1 syringe at the cecum and 1 syringe in the sigmoid colon. Up to 2 additional doses can be delivered at the discretion of the endoscopist up to a maximum of 4 total doses (max total dose = 80 ml of Solution B, also has 0 mg of L-Menthol).
  Arms: Placebo

SUMMARY:
The primary objective of this double-blinded, prospective, randomized placebo-controlled study is to evaluate for change in endoscopic adenoma detection rates (ADR) with the use of peppermint oil solution vs placebo application during colonoscopy. The investigators hypothesize that ADR will be increased with the use of the peppermint oil solution and thus further reduce the risk of colon cancer by means of colonoscopy.

DETAILED DESCRIPTION:
Adult subjects who are undergoing colonoscopy for primary colorectal cancer screening or surveillance. The study will be carried out as a prospective, double-blinded, fully-masked randomized controlled trial. Prior to the trial entry, the participant's labs and medical record will be reviewed in the electronic records system. If the subject meets inclusion/exclusion criteria, he or she will be consented at bedside prior undergoing their scheduled procedure and receive standard care as otherwise. Experimental and placebo solution ingredients will be serially numbered and randomized in a 1:1 ratio using a variable block strategy and provided by the institutional investigational pharmacy. Research staff will draw up experimental or placebo solution in 4 syringes with a total of 20mL in each solution.

The solutions are identical in appearance and endoscopic delivery. To prevent olfactory detection of the peppermint oil solution an essential oil diffuser will be used in all endoscopy rooms using the same oil as in the experimental solution. Endoscopists will be instructed to deliver the contents of one syringe sprayed via the endoscope in the cecum and one in the sigmoid colon. The contents of the other two syringes are to be delivered at the discretion of the endoscopist. After the procedure, endoscopists and study participants will be surveyed to determine if blinding was effective and to assess patient comfort levels, respectively. The primary and secondary end points will be determined on an intention to treat basis.

ELIGIBILITY:
Inclusion Criteria:

1. At least 50 years of age in Caucasians or 45 years of age in African-Americans.
2. Patients undergoing primary screening colonoscopy (either average risk or increased-risk) or surveillance colonoscopy after prior screening/surveillance colonoscopy.
3. Capable of understanding instructions, adhering to study schedules and requirements, and willing to provide informed consent.

Exclusion Criteria:

1. History of colectomy, partial or complete
2. Symptoms suggesting possible colorectal stenosis or cancer
3. Inflammatory bowel disease
4. Familial polyposis syndromes
5. History of, or current diagnosis of colorectal cancer
6. American Society of Anesthesia Physical Stats (ASA PS) score of IV or greater
7. Non-correctable coagulopathy
8. Currently receiving anti-thrombotic therapy, with an INR > 1.5
9. Poor prep, total BBPS score < 6, or any part of the colon < 2.
10. Patients with known allergy to peppermint oil or peppermint containing products.
11. Patients taking calcium channel blockers (Amlodipine, Nifedipine, Verapamil, Diltiazem, Dihydropyridine, Felodipine, etc).

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Wong, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Day1 - patients undergoing screening and surveillance colonoscopy are pre-screened to evaluate if they meet inclusion criteria.
  Once identified patient is approached by study personnel to determine their willingness. If willing to participate will undergo written consent for participation. Patients will be followed up by telephone for adverse reactions at 24-48 hr, one week and one month after colonoscopy.
Pre-assignment Details: Patients will be questioned regarding their allergy status specific to peppermint oil and this will be documented in the consent form and in the RedCap database. The patient must meet all inclusion and exclusion criteria and willing to participate in informed consent.
Groups:
- Placebo: Solution B) Placebo solution
  Ingredients:
  1. 0.4mL of Tween® 80 (i.e. Polysorbate 80) - this is a commonly used food additive that acts as a surfactant to bring the peppermint oil into solution
  2. 1L prepackage sterile water
  3. 2.6mL of undyed simethicone
     Instructions to prepare:
  4. Add tween and simethicone to sterile water. Then, shake vigorously.
  5. Once solution has settled, and patient has been randomized, draw 20mL of solution into a plastic syringe
  Placebo: During the colonoscopy the Endoscopists will be required to deliver intraluminally 1 syringe at the cecum and 1 syringe in the sigmoid colon. Up to 2 additional doses can be delivered at the discretion of the endoscopist up to a maximum of 4 total doses (max total dose =80 ml Solution B which contains 0 mg of L-Menthol).
- Peppermint Oil: Solution A) Peppermint oil solution (1.6% peppermint oil, which is 0.8% L-menthol)
  Ingredients:
  1. 16mL of peppermint oil (provided by the NowFoods® company)
  2. 0.4mL of Tween® 80 (i.e. Polysorbate 80) - this is a commonly used food additive that acts as a surfactant to bring the peppermint oil into solution
  3. 1L prepackage sterile water
  4. 2.6mL of undyed simethicone
  Peppermint Oil: During the colonoscopy the Endoscopists will be required to deliver intraluminally 1 syringe at the cecum and 1 syringe in the sigmoid colon. Up to 2 additional doses can be delivered at the discretion of the endoscopist up to a maximum of 4 total doses (max total dose = 640mg L-Menthol).
Period: Overall Study
Arm/Group | Placebo | Peppermint Oil
Started | 42 | 40
Completed | 38 | 37
Not Completed | 4 | 3
Not completed — Physician Decision | 4 | 3

BASELINE CHARACTERISTICS:
Population: The study protocol did not collect race or ethnicity.
Groups:
- Placebo: Solution B) Placebo solution
  Ingredients:
  1. 0.4mL of Tween® 80 (i.e. Polysorbate 80) - this is a commonly used food additive that acts as a surfactant to bring the peppermint oil into solution
  2. 1L prepackage sterile water
  3. 2.6mL of undyed simethicone
     Instructions to prepare:
  4. Add tween and simethicone to sterile water. Then, shake vigorously.
  5. Once solution has settled, and patient has been randomized, draw 20mL of solution into a plastic syringe
  Placebo: During the colonoscopy the Endoscopists will be required to deliver intraluminally 1 syringe at the cecum and 1 syringe in the sigmoid colon. Up to 2 additional doses can be delivered at the discretion of the endoscopist up to a maximum of 4 total doses (max total dose = 80 ml of Solution B ; with 0 mg of L-Methol).
- Total: Total of all reporting groups
Arm/Group | Placebo | Peppermint Oil | Total
Number analyzed (Participants) | 38 | 37 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 30 | 58
  >=65 years | 10 | 7 | 17
Age, Continuous [Median (Standard Deviation); unit: years] | 60.5 (6.75) | 67.73 (8.8) | 60.5 (7.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 25 | 46
  Male | 17 | 12 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38 | 37 | 75

OUTCOME MEASURES:

1. Primary Outcome: Adenoma Detection Rates
Description: Evaluate for changes in adenoma detection rates with the use of intraluminal peppermint oil application vs sterile water application during colonoscopy.
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Solution B) Placebo solution
  Ingredients:
  1. 0.4mL of Tween® 80 (i.e. Polysorbate 80) - this is a commonly used food additive that acts as a surfactant to bring the peppermint oil into solution
  2. 1L prepackage sterile water
  3. 2.6mL of undyed simethicone
     Instructions to prepare:
  4. Add tween and simethicone to sterile water. Then, shake vigorously.
  5. Once solution has settled, and patient has been randomized, draw 20mL of solution into a plastic syringe
  Placebo: During the colonoscopy the Endoscopists will be required to deliver intraluminally 1 syringe at the cecum and 1 syringe in the sigmoid colon. Up to 2 additional doses can be delivered at the discretion of the endoscopist up to a maximum of 4 total doses (max total dose = 80 ml of Solution B ; 0 mg of L-Menthol)
Arm/Group | Peppermint Oil | Placebo
Number analyzed (Participants) | 37 | 38
Participants
  Adenoma Detected "Yes" Yes Adenoma Detected | 19 | 20
  Adenoma Detected "No" | 18 | 18

2. Secondary Outcome: Polyp Detection Rates
Description: Evaluate for changes in Polyp detection rates.
Time Frame: 1 week .
Measure: Count of Participants; unit: Participants
Arm/Group | Peppermint Oil | Placebo
Number analyzed (Participants) | 37 | 38
Participants
  Polyp detected "Yes" | 30 | 29
  Polyp detected "No" | 7 | 9

3. Secondary Outcome: Procedure Time
Description: Evaluate for changes in total procedure time, cecal intubation time, and withdrawal time with the use of intraluminal peppermint oil application vs sterile water application during colonoscopy.
Time Frame: immediate
Population: Note that total procedure time was not collected
Measure: Median (Full Range); unit: minutes
Groups:
- Peppermint Oil: Solution A) Peppermint oil solution (1.6% peppermint oil, which is 0.8% L-menthol)
  Ingredients:
  1. 16mL of peppermint oil (provided by the NowFoods® company)
  2. 0.4mL of Tween® 80 (i.e. Polysorbate 80) - this is a commonly used food additive that acts as a surfactant to bring the peppermint oil into solution
  3. 1L prepackage sterile water
  4. 2.6mL of undyed simethicone
  Peppermint Oil: During the colonoscopy the Endoscopists will be required to deliver intraluminally 1 syringe at the cecum and 1 syringe in the sigmoid colon. Up to 2 additional doses can be delivered at the discretion of the endoscopist up to a maximum of 4 total doses (max total dose = 640mg L-Mentol).
Arm/Group | Peppermint Oil | Placebo
Number analyzed (Participants) | 37 | 38
minutes
  Cecal Intubation time in minutes | 12.4 [4.1 to 46.7] | 12.9 [3.9 to 22.8]
  Withdraw Time in minutes | 20.5 [6.1 to 31.2] | 17.2 [0.5 to 42.7]

4. Secondary Outcome: Advanced Adenoma Detection Rates
Description: Evaluate for changes in advanced adenoma detection rates with the use of intraluminal peppermint oil application vs placebo during coloscopy. Advanced adenoma will be define as an adenoma with significant villous features (>25%), size of 1.0 cm or more, high-grade dysplasia, or early invasive cancer.
Time Frame: 2 weeks
Population: The data was not entered in the database in a format that would allow it to be collated according to the definition above. Also, some subjects did show more than one advanced adenoma.
Measure: Number; unit: participants
Groups:
- Placebo: Solution B) Placebo solution
  Ingredients:
  1. 0.4mL of Tween® 80 (i.e. Polysorbate 80) - this is a commonly used food additive that acts as a surfactant to bring the peppermint oil into solution
  2. 1L prepackage sterile water
  3. 2.6mL of undyed simethicone
     Instructions to prepare:
  4. Add tween and simethicone to sterile water. Then, shake vigorously.
  5. Once solution has settled, and patient has been randomized, draw 20mL of solution into a plastic syringe
  Placebo: During the colonoscopy the Endoscopists will be required to deliver intraluminally 1 syringe at the cecum and 1 syringe in the sigmoid colon. Up to 2 additional doses can be delivered at the discretion of the endoscopist up to a maximum of 4 total doses (max total dose = 80 ml of Solution B, 0 mg of L-Menthol).
Arm/Group | Peppermint Oil | Placebo
Number analyzed (Participants) | 37 | 38
participants
  Tubular Adenoma | 19 | 19
  Tubulovillous Adenoma | 0 | 0
  Villous Adenoma | 0 | 0
  Serrated Adenoma | 1 | 4
  Cancer | 1 | 1
  No Adenoma | 18 | 18

5. Secondary Outcome: Cancer Detection Rates
Description: Evaluate for changes in cancer detection rates with the use of intraluminal peppermint oil application vs placebo during colonoscopy.
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Solution B) Placebo solution
  Ingredients:
  1. 0.4mL of Tween® 80 (i.e. Polysorbate 80) - this is a commonly used food additive that acts as a surfactant to bring the peppermint oil into solution
  2. 1L prepackage sterile water
  3. 2.6mL of undyed simethicone
     Instructions to prepare:
  4. Add tween and simethicone to sterile water. Then, shake vigorously.
  5. Once solution has settled, and patient has been randomized, draw 20mL of solution into a plastic syringe
  Placebo: During the colonoscopy the Endoscopists will be required to deliver intraluminally 1 syringe at the cecum and 1 syringe in the sigmoid colon. Up to 2 additional doses can be delivered at the discretion of the endoscopist up to a maximum of 4 total doses (max total dose = 80 ml of Solution B, 0 mg of L-Methol).
Arm/Group | Peppermint Oil | Placebo
Number analyzed (Participants) | 37 | 38
Participants
  Cancer detected "Yes" | 1 | 1
  Cancer detected "No" | 36 | 37

6. Secondary Outcome: Patient Comfort Level Recorded on Post-procedure Survey
Description: Evaluate for changes in reported patient comfort levels with the use of intraluminal peppermint oil application vs placebo during colonoscopy.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Solution B) Placebo solution
  Ingredients:
  1. 0.4mL of Tween® 80 (i.e. Polysorbate 80) - this is a commonly used food additive that acts as a surfactant to bring the peppermint oil into solution
  2. 1L prepackage sterile water
  3. 2.6mL of undyed simethicone
     Instructions to prepare:
  4. Add tween and simethicone to sterile water. Then, shake vigorously.
  5. Once solution has settled, and patient has been randomized, draw 20mL of solution into a plastic syringe
  Placebo: During the colonoscopy the Endoscopists will be required to deliver intraluminally 1 syringe at the cecum and 1 syringe in the sigmoid colon. Up to 2 additional doses can be delivered at the discretion of the endoscopist up to a maximum of 4 total doses (max total dose = 80 ml of Solution B; 0mg of L- Menthol).
Arm/Group | Peppermint Oil | Placebo
Number analyzed (Participants) | 37 | 38
Participants
  No Discomfort | 17 | 19
  Slight Discomfort | 15 | 15
  Moderate(bothersome) | 5 | 1
  Severe | 0 | 0
  Not available | 0 | 3

ADVERSE EVENTS:
Time Frame: Patients were assessed day one after procedure, 24-48 after, one week and one month after procedure
Description: patients were assessed and graded by AE definitions adapted from the National Cancer Institute Common Terminology Criteria for Adverse Events. Grades 1 through 5. Data was stored in RedCap.
Groups:
- Peppermint Oil: Solution A) Peppermint oil solution (1.6% peppermint oil, which is 0.8% L-menthol)
  Ingredients:
  1. 16mL of peppermint oil (provided by the NowFoods® company)
  2. 0.4mL of Tween® 80 (i.e. Polysorbate 80) - this is a commonly used food additive that acts as a surfactant to bring the peppermint oil into solution
  3. 1L prepackage sterile water
  4. 2.6mL of undyed simethicone
  Peppermint Oil: During the colonoscopy the Endoscopists will be required to deliver intraluminally 1 syringe at the cecum and 1 syringe in the sigmoid colon. Up to 2 additional doses can be delivered at the discretion of the endoscopist up to a maximum of 4 total doses (max total dose = 640mg Placebo).
- Placebo: Solution B) Placebo solution
  Ingredients:
  1. 0.4mL of Tween® 80 (i.e. Polysorbate 80) - this is a commonly used food additive that acts as a surfactant to bring the peppermint oil into solution
  2. 1L prepackage sterile water
  3. 2.6mL of undyed simethicone
     Instructions to prepare:
  4. Add tween and simethicone to sterile water. Then, shake vigorously.
  5. Once solution has settled, and patient has been randomized, draw 20mL of solution into a plastic syringe
  Placebo: During the colonoscopy the Endoscopists will be required to deliver intraluminally 1 syringe at the cecum and 1 syringe in the sigmoid colon. Up to 2 additional doses can be delivered at the discretion of the endoscopist up to a maximum of 4 total doses (max total dose = 640mg Placebo).
Arm/Group | Peppermint Oil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/38
Other Adverse Events (participants affected / at risk) | 7/37 | 8/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peppermint Oil (N=37) | Placebo (N=38)
bloating and cramping (Gastrointestinal disorders) | 1 (1) | 4 (4)
Loss of appetite (Gastrointestinal disorders) | 1 (1) | 0 (0)
cramping (Gastrointestinal disorders) | 1 (1) | 2 (2)
bloating (Gastrointestinal disorders) | 2 (2) | 0 (0)
bumps (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
constipation and bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1)
hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-21): https://cdn.clinicaltrials.gov/large-docs/48/NCT02588248/Prot_SAP_002.pdf